CLINICAL TRIAL: NCT00252876
Title: An Open-Label, Multi-Centre and Long-Term Extension Study to Evaluate the Safety and Tolerability of Oral Tesaglitazar 1 mg in Patients With Type 2 Diabetes Mellitus.
Brief Title: GALLEX 1 - Long Term Extension Study in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6160C00038; GALLEX 1
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar

INTERVENTIONS:
Drug: tesaglitazar

SUMMARY:
This is a 107-week open-label, multi-center long-term extension study from GALLANT studies 2/22, 5, 7, 8 and 14 to monitor the safety and tolerability of oral tesaglitazar 1 mg in patients with type 2 diabetes during up to 104 weeks of treatment. The total duration, including treatment and follow-up, is 107 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=18 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Completed the last two visits of randomized treatment period in GALLANT 2/22, 5, 7, 8 or 14 studies.

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Previous enrollment in this long-term extension study
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2005-03; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory variables, physical examination, cardiac evaluation, hypoglycemic events, electrocardiogram, vital signs (blood pressure and pulse), body weight

SECONDARY OUTCOMES:
Pharmacodynamic: fasting plasma glucose, glycosylated hemoglobin A1c, lipid variables (triglyceride, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol)
Responder rates and proportion of patients on tesaglitazar who reach pre-specified target levels for triglyceride, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and non-high-density lipoprotein cholesterol
C-reactive protein
Central obesity (waist circumference, hip circumference, waist/hip ratio)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (277):
- United States (58):
  - Research Site, Birmingham, Alabama
  - Research Site, Columbiana, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Carlisle, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Chula Vista, California
  - Research Site, Escondido, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Pasadena, California
  - Research Site, Redondo Beach, California
  - Research Site, Sacramento, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Brunswick, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Evansville, Indiana
  - Research Site, Witchita, Kansas
  - Research Site, Bossier City, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Hamilton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, White Plains, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Simpsonville, South Carolina
  - Research Site, Morristown, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Burke, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Menomonee Falls, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Morón, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Rosario
  - Research Site, Salta - Salta
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Cairns
  - Research Site, Geelong
  - Research Site, Melbourne
  - Research Site, Perth
  - Research Site, Sydney
  - Research Site, Tasmania
- Brazil (6):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (22):
  - Research Site, Calgary, Alberta
  - Research Site, Coquitlam, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bolton, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Hastings, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Napanee, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Smith Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chomedey-Laval, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (9):
  - Research Site, Brno
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Příbram
  - Research Site, Semily
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
- Estonia (5):
  - Research Site, Paide
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
  - Research Site, Viljandi
- Finland (17):
  - Research Site, Hämeenlinna
  - Research Site, Helsinki
  - Research Site, Imatra
  - Research Site, Jakobstad
  - Research Site, Joensuu
  - Research Site, Kokkola
  - Research Site, Kouvola
  - Research Site, Kuopio
  - Research Site, Lahti
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Salo
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Turku
  - Research Site, Vaasa
  - Research Site, Vantaa
- Greece (2):
  - Research Site, Athens
  - Research Site, Piraeus
- Research Site, Hong Kong, Hong Kong
- Hungary (8):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Siófok
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Bangalore
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, New Delhi
- Indonesia (2):
  - Research Site, Jakarta
  - Research Site, Malang
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Rishon LeZiyyon
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (17):
  - Research Site, Arenzano
  - Research Site, Chiavari (GE)
  - Research Site, Chieri
  - Research Site, Florence
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Monteccio Emilia
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Pescara
  - Research Site, Piacenza
  - Research Site, Pistoia
  - Research Site, Reggio Calabria
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Scandiano
  - Research Site, Udine
- Latvia (7):
  - Research Site, Daugavpils
  - Research Site, Jēkabpils
  - Research Site, Madona
  - Research Site, Riga
  - Research Site, Sigulda
  - Research Site, Talsi
  - Research Site, Valmiera
- Research Site, Vilnius, Lithuania
- Malaysia (3):
  - Research Site, Kubang Kerian, Kota Bharu
  - Research Site, George Town
  - Research Site, Kuala Lumpur
- Netherlands (10):
  - Research Site, Beek en Donk
  - Research Site, Bennebroek
  - Research Site, Deurne
  - Research Site, Huizen
  - Research Site, Losser
  - Research Site, Nijverdal
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, The Hague
- Philippines (6):
  - Research Site, Cebu City
  - Research Site, Makati
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
  - Research Site, Quezon City
- Poland (17):
  - Research Site, Katowice, Ochojec
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Toruñ
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zielona Góra
- Portugal (5):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Elvas
  - Research Site, Lisbon
  - Research Site, Portalegre
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Research Site, Belgrade, Serbia and Montenegro
- Research Site, Singapore, Singapore
- Slovakia (10):
  - Research Site, Dolný Kubín
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Ľubochňa
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Šahy
  - Research Site, Trenčín
  - Research Site, Veľký Meder
  - Research Site, Žilina
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, Chatsworth
  - Research Site, Durban
  - Research Site, Gauteng
  - Research Site, Johannesburg
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Switzerland (5):
  - Research Site, Bern
  - Research Site, Ilanz
  - Research Site, Lausanne
  - Research Site, Monthey
  - Research Site, Zurich
- United Kingdom (25):
  - Research Site, Aberdeen
  - Research Site, Atherstone
  - Research Site, Ayr
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Berks
  - Research Site, Birmingham
  - Research Site, Bolton
  - Research Site, Bucks
  - Research Site, Cardiff
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Plymouth
  - Research Site, Radstock
  - Research Site, Shrewsbury
  - Research Site, Surrey
  - Research Site, West Bromwich
  - Research Site, Wiltshire
  - Research Site, Wrexham
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City